CLINICAL TRIAL: NCT00145756
Title: China Salt Substitute Study-A Randomised Trial to Determine the Long-Term Effects of a Low Sodium, High Potassium Salt Substitute on Blood Pressure Among High-Risk Individuals in Northern China
Brief Title: China Salt Substitute Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Fu Wai Cardiovascular Institute and Hospital (Unknown); University of Auckland, New Zealand (Other); James Cook University, Queensland, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CSSS
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Sodium Chloride; Blood Pressure; Cardiovascular Diseases; Clinical Trial
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

INTERVENTIONS:
Drug: low sodium high potassium salt substitute

SUMMARY:
Cardiovascular disease is a leading cause of death and disability worldwide, and blood pressure is a leading determinant of this risk. To date, strategies for blood pressure lowering have focused on drug treatment but dietary interventions such as reducing sodium intake and increasing potassium intake may also be effective. Such interventions may be particularly suitable for low- and middle-income countries in which significant dietary changes may be more easily achieved. This study will test the effect of a salt substitute on blood pressure, among individuals at high-risk from cardiovascular disease in Northern China.

DETAILED DESCRIPTION:
This randomised trial will clearly identify whether a low-sodium, high-potassium salt-substitute is a feasible means of lowering blood pressure in high-risk individuals in rural China. The randomised design and the large size (n=600) will ensure that the results are reliable and precise. The 12-month duration will address the long-term practicability of the intervention strategy. The study is being conducted because salt-substitute-based blood pressure lowering may be particularly appropriate for rural populations in low- and middle-income countries. First, sodium intake is often very high. Second, the salt-substitute can be easily incorporated into the diet because most food is prepared and eaten at home. Third, the intervention can be provided at very low cost.

Comparisions: Low sodium high potassium salt (65% sodium chloride, 25% potassium chloride, 10% magnesium sulphate) compared to normal salt (100% sodium chloride).

ELIGIBILITY:
Inclusion Criteria:

Participant inclusion will be based upon the presence of:

* A doctor-confirmed high risk of future vascular disease defined as a history of any one of:

  * Stroke or transient ischaemic attack
  * Hospitalisation for management of any acute coronary syndrome
  * Surgery or angioplasty for peripheral vascular disease
  * Treated diabetes and age 55 years or older
  * Systolic blood pressure >160mmHg
* Estimated daily sodium intake of 260mmol/24hrs (about 15g/24hrs of NaCl) or above and expectation that at least 50% of daily dietary salt intake can be replaced with the salt-substitute. This will be estimated through interview of the potential participant and the individual responsible for daily food preparation (if this is not the patient) using a structured questionnaire.
* Provision of informed consent

Exclusion Criteria:

Potential participants will be excluded if:

* they are on potassium-sparing medication
* there is an established history of significant renal impairment that would preclude the use of the salt-substitute in the opinion of the responsible physician.
* there is any reason why either the salt-substitute or normal salt are definitely indicated or definitely contra-indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-05; Study Completion 2005-09

PRIMARY OUTCOMES:
Clinical blood pressure

SECONDARY OUTCOMES:
Spot urine sodium and potassium levels
Food taste
Preferred level of saltiness

CONTACTS AND LOCATIONS:
Overall Officials: Bruce C Neal, PhD, Principal Investigator — The George Institute; Yangfeng Wu, PhD, Principal Investigator — Fu Wai Cardiovascular Institute, Beijing, China; Rachel Huxley, PhD, Principal Investigator — The George Institute; John Prescott, PhD, Principal Investigator — James Cook University, Queensland, Australia
Locations (6):
- China (6):
  - The Institute for Medical Science of Mudangjiang, Mudanjiang, Heilongjiang
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The People's Hospital of YuXian, Yangquan, Shanxi
  - The Health Center of Fengbo,ShunYi District, Beijing
  - The Health Center of YingHai, DaXing District, Beijing
  - The First Affiliated Hospital of Medical College of China's people Armed Police Force, Tianjin

REFERENCES:
- [Derived] Kissock K, Neal B, Yuan Y, Sundstrom J, Jonsson H, Rodgers A, Wang N, Huang L, Wu Y. Consistency of Blood Pressure Response to Potassium-Enriched Salt in the China Salt Substitute Study. Hypertension. 2026 Jan;83(1):167-176. doi: 10.1161/HYPERTENSIONAHA.125.24723. Epub 2025 Nov 20. PMID 41263071